CLINICAL TRIAL: NCT04565210
Title: Effects of Oriental Music oN Preterm InfAnts: A Randomized Controlled Trial. (OMNIA Trial)
Brief Title: Effects of Oriental Music on Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBS-2020-0284
Record Dates: First submitted 2020-09-07; First posted 2020-09-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-10

CONDITIONS: Premature; Behavior, Child
Keywords: Music therapy; Premature infant; Heart rate variability; Behavior state
MeSH Terms: conditions — Premature Birth; Child Behavior | interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oriental music (Experimental): Infants assigned to this group will be exposed to oriental music.
  Interventions: Other: Music exposure
- Western music (Active Comparator): Infants assigned to this group will be exposed to western music.
  Interventions: Other: Music exposure
- Silence / control (Placebo Comparator): Infants assigned to this group will be exposed to the same protocol but using a track of silence.
  Interventions: Other: Silence

INTERVENTIONS:
Other: Music exposure — Participants will be offered individual sessions of music. They will be exposed for 10 minutes per day, 3 days per week for a period of 2 weeks using a headphone.
  Arms: Oriental music; Western music
Other: Silence — Participants in this group will be offered individual silence session for 10 minutes per day, 3 days per week for a period of 2 weeks using a headphone.
  Other Names: No music
  Arms: Silence / control

SUMMARY:
The goal of this study is to explore the effect of oriental music on premature infants' physiological and behavioral parameters during their hospital stay in the NICU.

DETAILED DESCRIPTION:
Music exposure during care of preterm infants is the subject of increasing research. Many studies have shown positive impact of music exposure such as classical western music, lullabies or Quran on pain and physiological parameters of preterm infants in a neonatal intensive care unit (NICU) setting. No such study have explored the effect of oriental music which is the main popular music listened to in the Levant and Middle East and North Afrika (MENA) region.

We aim in this study to find out if the oriental music exposure in preterm infants improves babies' heart rate variability, physiological parameters and behavior state during their NICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable infants born between 28 and 366/7 weeks of gestation and ≥31 weeks Post Menstrual Age (PMA).
* Infants planned to stay in the NICU for at least 2 weeks at the time of enrollment.

Exclusion Criteria:

* Congenital anomaly affecting heart rate and hearing, significant brain insult (such as severe or moderate hypoxic ischemic encephalopathy, intraventricular hemorrhage (IVH) grade 3 or 4 or periventricular leukomalacia) that might affect the neurodevelopmental outcome.
* Receiving medications that might interfere with heart rate and reaction to music exposure such as midazolam or morphine.

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 3 years
  It consists of changes in the time intervals between consecutive heartbeats called inter-beat intervals (RR).

SECONDARY OUTCOMES:
Mean Respiratory rate | 3 years
  The respiratory rate will be retrieved from bedside monitors.
Oxygen Saturation | 3 years
  The oxygen saturation will be retrieved from bedside monitors.
Behavioral state | 3 years
  The behavioral score will be assessed using a 7- point score by a certified nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No